CLINICAL TRIAL: NCT02665351
Title: A Phase 2, Pilot, Open-label, Randomized Study of the Antiviral Activity, Safety, and Tolerability of Intravenous Peramivir in Adult Hospitalized Subjects With Confirmed Influenza Infection
Brief Title: Peramivir Treatment Response in Adults Hospitalized for Influenza-associated Lower Respiratory Tract Infections
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Collaborators: BioCryst Pharmaceuticals (Industry)
Responsible Party: Principal Investigator, Prof David Shu Cheong Hui, Professor, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Peramivir in adult influenza_1
Record Dates: First submitted 2016-01-22; First posted 2016-01-27 (Estimated); Last update posted 2016-01-29 (Estimated); Status verified 2016-01

CONDITIONS: Influenza
MeSH Terms: conditions — Influenza, Human | interventions — peramivir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Peramivir 300mg Q12H (Active Comparator): Peramivir 300 mg, administered intravenously, twice daily (every 12 hours)
  Interventions: Drug: Peramivir
- Peramivir 600mg Q24H (Active Comparator): Peramivir 600 mg, administered intravenously, once daily (every 24 hrs)
  Interventions: Drug: Peramivir

INTERVENTIONS:
Drug: Peramivir — The two regimens of Peramivir were compared
  Other Names: intravenous neuraminidase inhibitor

SUMMARY:
Peramivir is the first intravenous neuraminidase inhibitor (NAI) available for treatment of uncomplicated influenza in adults. Data from placebo-controlled trials in outpatients have shown antiviral efficacy, safety, and tolerability. Although the unmet need for intravenous therapy lies mainly with patients hospitalized with complicated diseases, such data are limited because of feasibility and ethical considerations for placebo-controlled studies.

In this study, the investigators aimed to examine more specifically treatment effects of peramivir in adults hospitalized with influenza-associated lower respiratory tract complications (LRTC). Such findings may have important implications on clinical management.

DETAILED DESCRIPTION:
The primary objective was to assess the virologic response of peramivir in influenza-associated lower respiratory tract complications (LRTC). The secondary objective was to assess safety and tolerability. Adults confirmed with influenza by polymerase chain reaction (PCR) and/or immunofluorescence assays during the seasonal peaks of 2011-2014 were assessed for eligibility. Consented individuals were randomized to receive either peramivir 600mg every 24 hourly or 300mg every 12 hourly for 5 days. In subjects not achieving clinical resolution by day 5, the same regimen could be continued until day 10 (virologic results unknown to clinicians).Renal-dosage adjustment, if required, was performed according to protocol.

The study's primary endpoint was change in influenza RNA load over time. The secondary endpoints were viral shedding indicated by culture and RNA negativity at day 5, and drug tolerability.

Additionally, a priori comparisons of these endpoints with historical controls treated with standard courses of oral oseltamivir (75mg bid for 5 days) in the same clinical settings were performed.

ELIGIBILITY:
Inclusion Criteria:

* symptoms/signs of influenza, and
* confirmation of lower respiratory tract infection (e.g. radiographic pneumonia, dyspnea caused by acute exacerbation of underlying airway diseases, bronchitis, or combinations).

Exclusion Criteria:

* late presentation >1 week from onset,
* hemodynamic instability,
* hepatic/renal failure,
* dialysis,
* immunosuppression (e.g. transplant, chemotherapy), and
* pregnancy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2011-02; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
change in influenza RNA load | 5 days
  5-10 days

SECONDARY OUTCOMES:
viral shedding indicated by PCR and culture negativity | 5 days

CONTACTS AND LOCATIONS:
Overall Officials: Nelson Lee, Principal Investigator — Chinese University of Hong Kong
Locations (1):
- Prince of Wales Hospital, Hong Kong, Hong Kong, China

IPD SHARING:
Plan to Share IPD: No